CLINICAL TRIAL: NCT06309550
Title: Provocative Tests for Diagnosing and Phenotyping Heart Failure With Preserved Ejection Fraction
Brief Title: Provocative Tests for HFpEF
Acronym: TEST-PEF
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09W002
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: exercise test — exercise test

SUMMARY:
Diagnosing heart failure with preserved ejection fraction (HFpEF) in patients complaining exertional breathlessness can be challenging: diagnostic algorithms and scores have low sensitivity, and ageing-associated comorbidities can complicate the interpretation of symptoms. Thus, exercise right heart catheterization (RHC) or invasive cardiopulmonary exercise test (iCPET) have been advocated as gold-standard methods for HFpEF diagnosis. However, exercise RHC and iCPET are still not widely standardized methods, with results mainly coming from US cohorts (that may differ from Italian cohorts), and other provocative tests (e.g. non-invasive CPET, passive leg raising) may offer complementary diagnostic information.

ELIGIBILITY:
Inclusion Criteria:

* dyspnea

Exclusion Criteria:

* known HFpEF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients referred to the Dyspnea and Pulmonary Hypertension Center for suspicion of HF, PH or unexplained dyspnea
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
  Incidence of mortality
Hospitalization for heart failure | 5 years
  Incidence of hospitalization for heart failure
Atrial fibrillation | 5 years
  Incidence of atrial fibrillation

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Luca IRCCS Istituto Auxologico Italiano, Milan, Italy